CLINICAL TRIAL: NCT02301026
Title: A Non-interventional Study of Diafer (5% Iron Isomaltoside 1000) Administered According to Standard Hospital Practice and Product Labelling in Subjects With Chronic Kidney Disease on Haemodialysis for Treatment of Iron Deficiency
Brief Title: A Non-interventional Study of Diafer in Subjects With CKD on Haemodialysis for Treatment of Iron Deficiency
Acronym: DINO
Status: Completed | Type: Observational
Sponsor: Pharmacosmos A/S (Industry)
Collaborators: BioStata (Industry)
Responsible Party: Sponsor
Other Study IDs: Diafer-NIS-06
Record Dates: First submitted 2014-10-13; First posted 2014-11-25 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-04

CONDITIONS: Anaemia in Chronic Kidney Disease
MeSH Terms: interventions — iron isomaltoside 1000

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: 5% Iron Isomaltoside 1000 — Administered according to local routines and product labeling in doses at the doctors discretion
  Other Names: Diafer®

SUMMARY:
The purpose of the study is to monitor initiated Diafer® therapy administered according to hospital practice and the product labeling in routine clinical practice in haemodialysis patients with Chronic Kidney Disease.

DETAILED DESCRIPTION:
Parenteral iron is the iron treatment of choice for haemodialysis (HD) patients with Chronic Kidney Disease (CKD), who may suffer from absolute iron deficiency due to continuous blood losses and/or functional iron deficiency due to erythropoiesis stimulating agent treatment or impaired release from iron stores.

Much evidence indicates that adequate iron supply is necessary to achieve optimal responses to ESAs and thereby potentially avoid ESA induced ADRs.

Pharmacosmos has been working with dialysis providers for many years and identified a medical need for a new safe and cost-effective low dose intravenous (IV) iron that can be administered frequently. Diafer® is a new low dose iron formulation based on iron isomaltoside 1000, with doses restricted to maximum 200 mg iron pr. injection. No test dose is needed and Diafer® may be administered as a push injection.

The primary objective of the study is to monitor initiated Diafer® therapy administered according to hospital practice and the product labeling in routine clinical practice in HD patients with CKD. The scientific rationale being to fulfil a need for systematic information/auditing on applied practice including long term experience with the use of IV iron in the HD setting. This information will provide an evidence base for optimised treatment procedures.

ELIGIBILITY:
Inclusion Criteria:

* HD patients ≥ 18 years of age in a stable phase of CKD as judged by the investigator
* Patients must have been on HD > 3 months
* Patients must have received at least one dose of iron sucrose treatment within the last 6 months

Exclusion Criteria:

* Diafer® contraindications
* Patient not able to give informed consent
* Significant disease not related to CKD and likely to impact study results as evaluated by investigator
* Inability to estimate retrospective baseline data
* Planned change of iron dosing protocol or routines around iron administration during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients ≥ 18 years of age with chronic kidney disease (CKD) who have been on HD > 3 months and have received at least one dose of iron sucrose treatment within the last 6 months while being on dialysis.
Sampling Method: Non-Probability Sample
Enrollment: 209 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2016-12-09 (Actual); Study Completion 2016-12-09 (Actual)

PRIMARY OUTCOMES:
Hb (Change in Hb compared to baseline at 3 months intervals) | 12 month
  Change in Hb compared to baseline at 3 months intervals

SECONDARY OUTCOMES:
Adverse drug reactions | 12 month
Adverse Events | 12 month
  AEs of special interest defined as hypersensitivity symptoms such as urticaria, oedema, bronchospasm, hypotension, cardiorespiratory arrest, syncope, unresponsiveness or loss of consciousness at pre-specified time points in relation to administration of study drug
ESA (use of ESA and dose) | 12 month
  Use of ESA and dose
Blood Transfusion (Number of blood transfusions) | 12 month
  Number of blood transfusions
IV iron dose (Total needed dose) | 12 month
  Total needed dose

OTHER OUTCOMES:
Nurse hours (time spend per treatment) | 12 month
  Nurse time spend per treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sylvia Simon, Study Chair — Pharmacosmos A/S
Locations (2):
- Heleneholmsdialysen, Malmo, Sweden
- Morriston Hospital, Renal Department, Swansea, Wales, United Kingdom

REFERENCES:
- [Derived] Mikhail AI, Schon S, Simon S, Brown C, Hegbrant JBA, Jensen G, Moore J, Lundberg LDI. A prospective observational study of iron isomaltoside in haemodialysis patients with chronic kidney disease treated for iron deficiency (DINO). BMC Nephrol. 2019 Jan 10;20(1):13. doi: 10.1186/s12882-018-1159-z. PMID 30630452